CLINICAL TRIAL: NCT00717860
Title: A Multicenter, Double-Blind, Comparative Study of MK0991 (Caspofungin) Versus Micafungin in Adult Japanese Patients With Deep-seated Candida or Aspergillus Infections
Brief Title: A Clinical Study of MK0991 (Caspofungin) in Japanese Patients With Deep-seated Candida or Aspergillus Infections (0991-062)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0991-062; 2008_013
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Caspofungin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Caspofungin (Experimental): caspofungin acetate (MK0991)
  Interventions: Drug: caspofungin acetate
- Micafungin (Active Comparator): Micafungin sodium
  Interventions: Drug: Comparator: Micafungin sodium

INTERVENTIONS:
Drug: caspofungin acetate — Caspofungin acetate (50 mg/day for participants with esophageal candidiasis and 50 mg/day for participants with invasive candidiasis or aspergillosis after a 70 mg loading dose on Day 1), once daily intravenously (IV) for 1-4 weeks for esophageal candidiasis, 2-8 weeks for invasive candidiasis, 2-12 weeks for aspergillosis.
  Arms: Caspofungin
Drug: Comparator: Micafungin sodium — Micafungin sodium 150 mg/day, once daily IV, for 1-4 weeks for esophageal candidiasis, 2-8 weeks for invasive candidiasis, 2-12 weeks for aspergillosis.
  Arms: Micafungin

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of MK0991 in patients with deep-seated mycoses.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Patients In Whom A Causative Fungus Is Detected Before Treatment With The Study Drug Or Patients With Strongly Suspected Deep-Seated Fungal Infection Due To Candida species (Spp.) Or Aspergillus Spp.

Exclusion Criteria:

* Patients With Mycoses Other Than Ones Due To Candida Spp. Or Aspergillus Spp.
* Patients Who Will Receive Other Systemic Antifungal Agents For The First Time In Screening Period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kohno S, Izumikawa K, Yoshida M, Takesue Y, Oka S, Kamei K, Miyazaki Y, Yoshinari T, Kartsonis NA, Niki Y. A double-blind comparative study of the safety and efficacy of caspofungin versus micafungin in the treatment of candidiasis and aspergillosis. Eur J Clin Microbiol Infect Dis. 2013 Mar;32(3):387-97. doi: 10.1007/s10096-012-1754-z. Epub 2012 Oct 3. PMID 23052987

RESULTS

PARTICIPANT FLOW:
Groups:
- Caspofungin: Caspofungin acetate (50 mg/day for participants with esophageal candidiasis and 50 mg/day for participants with invasive candidiasis or aspergillosis after a 70 mg loading dose on Day 1), once daily intravenously (IV) for 1-4 weeks for esophageal candidiasis, 2-8 weeks for invasive candidiasis, 2-12 weeks for aspergillosis.
- Micafungin: Micafungin sodium 150 mg/day, once daily IV for 1-4 weeks for esophageal candidiasis, 2-8 weeks for invasive candidiasis, 2-12 weeks for aspergillosis.
Period: Overall Study
Arm/Group | Caspofungin | Micafungin
Started | 61 | 60
Completed | 34 | 32
Not Completed | 27 | 28
Not completed — Clinical adverse experience | 5 | 9
Not completed — Laboratory adverse experience | 2 | 2
Not completed — Lack of Efficacy | 7 | 13
Not completed — Discontinued for other reason | 6 | 1
Not completed — Withdrew consent | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caspofungin | Micafungin | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (11.2) | 69.3 (9.0) | 69.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 50 | 46 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Significant Drug-related Adverse Experience
Description: A significant drug-related adverse experience was defined as a serious drug-related adverse experience or a drug-related adverse experience leading to study therapy discontinuation.
Time Frame: 1-4 weeks for esophageal candidiasis, 2-8 weeks for invasive candidiasis, 2-12 weeks for aspergillosis
Population: All Participants as Treated (APaT) population.
Measure: Number; unit: Participants
Arm/Group | Caspofungin | Micafungin
Number analyzed (Participants) | 60 | 60
Participants | 3 | 6

2. Secondary Outcome: Number of Participants With a Specific Safety Finding
Description: A specific safety finding was defined as a drug-related adverse experience, a serious drug-related adverse experience, or a drug-related adverse experience leading to study therapy discontinuation.
Time Frame: 1-4 weeks for esophageal candidiasis, 2-8 weeks for invasive candidiasis, 2-12 weeks for aspergillosis
Population: APaT population.
Measure: Number; unit: Participants
Arm/Group | Caspofungin | Micafungin
Number analyzed (Participants) | 60 | 60
Participants
  Drug-related adverse experience | 23 | 25
  Serious drug-related adverse experience | 0 | 2
  Discontinued by drug-related adverse experience | 3 | 6

3. Secondary Outcome: Number of Participants With Favorable Overall Response at the End of Study Therapy
Description: Favorable overall response for each infection category of deep-seated fungal infections was based on the determination of the Independent Efficacy Assessment Committee.
Time Frame: 1-4 weeks for esophageal candidiasis, 2-8 weeks for invasive candidiasis, 2-12 weeks for aspergillosis
Population: Per Protocol Set (PPS) population.
Measure: Number; unit: Participants
Arm/Group | Caspofungin | Micafungin
Number analyzed (Participants) | 44 | 41
Participants
  Esophageal candidiasis (n=6, n=6) | 6 | 5
  Invasive candidiasis (n=3, n=1) | 3 | 1
  Aspergillosis (n=30, n=33) | 14 | 14

ADVERSE EVENTS:
Arm/Group | Caspofungin | Micafungin
Serious Adverse Events (participants affected / at risk) | 12/60 | 14/60
Other Adverse Events (participants affected / at risk) | 44/60 | 40/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin (N=60) | Micafungin (N=60)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 3 (3) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peritoneal mesothelioma malignant advanced (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caspofungin (N=60) | Micafungin (N=60)
Constipation (Gastrointestinal disorders) | 6 (7) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 7 (7)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (3)
Injection site pain (General disorders) | 4 (4) | 5 (7)
Malaise (General disorders) | 4 (6) | 4 (4)
Oedema (General disorders) | 4 (4) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 4 (6)
Nasopharyngitis (Infections and infestations) | 4 (4) | 5 (8)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Alanine aminotransferase increased (Investigations) | 6 (8) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 9 (12) | 6 (7)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 9 (9)
Blood glucose increased (Investigations) | 7 (7) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 4 (5) | 4 (4)
Blood potassium decreased (Investigations) | 6 (6) | 1 (1)
Blood potassium increased (Investigations) | 3 (3) | 5 (5)
Blood pressure increased (Investigations) | 3 (8) | 4 (4)
C-reactive protein increased (Investigations) | 5 (5) | 4 (4)
Eosinophil count increased (Investigations) | 3 (3) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 4 (4)
Whtie blood cell count increased (Investigations) | 2 (2) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
Headache (Nervous system disorders) | 6 (7) | 5 (9)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.